CLINICAL TRIAL: NCT06520176
Title: A Prospective, Multicenter, Randomized Controlled Study of Etoposide, Cytarabine Combined With Pegfilgrastim vs. Cyclophosphamide Combined With G-CSF for Hematopoietic Stem Cell Mobilization in Newly Diagnosed Multiple Myeloma Patients
Brief Title: Comparison Study of EAP and CG Regimens for Mobilizing Hematopoietic Stem Cells in Multiple Myeloma Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Affiliated People's Hospital of Ningbo University (Other Government)
Collaborators: First Affiliated Hospital of Zhejiang University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); The Central Hospital of Lishui City (Other); Jinhua People's Hospital (Other); Shaoxing People's Hospital (Other); Shaoxing Second Hospital (Other); Zhejiang Provincial Tongde Hospital (Other); Taizhou Hospital (Other); Dongyang People's Hospital (Other); Affiliated Hospital of Jiaxing University (Other); Huizhou Municipal Central Hospital (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Ningbo Medical Center Lihuili Hospital (Other Government); Jinhua Municipal Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-060
Record Dates: First submitted 2024-07-20; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Multiple Myeloma; Hematopoietic Stem Cell Mobilization
Keywords: Multiple Myeloma; Etoposide; Cytarabine; PEG-rhG-CSF; Hematopoietic Stem Cell Mobilization
MeSH Terms: conditions — Multiple Myeloma | interventions — Etoposide; Cytarabine; pegfilgrastim; pegylated granulocyte colony-stimulating factor; Cyclophosphamide; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, two-arm, multicenter, exploratory study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EAP regimen group (Experimental): 66 subjects will be enrolled into the EAP regimen group. EAP regimen is the combination of etoposide, cytarabine and PEG-rhG-CSF.
  Interventions: Drug: Etoposide; Drug: Cytarabine; Drug: Pegfilgrastim; Drug: G-CSF
- CG regimen group (Active Comparator): 33 subjects will be enrolled into the CG regimen group. CG regimen is the combination of cyclophosphamide and G-CSF.
  Interventions: Drug: Cyclophosphamide; Drug: G-CSF

INTERVENTIONS:
Drug: Etoposide — Day 1~Day 2: 75mg/m^2
  Other Names: VP-16
  Arms: EAP regimen group
Drug: Cytarabine — Day 1~Day 2: 200g/m^2, q12h
  Other Names: Ara-C
  Arms: EAP regimen group
Drug: Pegfilgrastim — Day 6: 6mg
  Other Names: PEG-rhG-CSF
  Arms: EAP regimen group
Drug: Cyclophosphamide — Day 1~Day 2: 1～2g/m^2
  Other Names: Cy
  Arms: CG regimen group
Drug: G-CSF — Subcutaneous injection at dose 5ug/kg, from day 6 until the end of mobilization.
  Other Names: Granulocyte Colony Stimulating Factor
  Arms: CG regimen group
Drug: G-CSF — Starting from the 9th day, if the white blood cell count is less than 20,000/μL, administer G-CSF at a dose of 5μg/kg by subcutaneous injection until the collection is completed.
  Other Names: Granulocyte Colony Stimulating Factor
  Arms: EAP regimen group

SUMMARY:
This is a prospective, randomized, two-arm, multicenter, exploratory study aimed at evaluating the efficacy and safety of the combination of etoposide, cytarabine and Pegfilgrastim (EAP regimen) for mobilizing hematopoietic stem cells in patients with newly diagnosed multiple myeloma (NDMM). A total of 99 NDMM patients will be enrolled and randomly assigned to receive either the EAP regimen or the GC regimen (cyclophosphamide+ G-CSF) to mobilize hematopoietic stem cells. Subsequently, the mobilization effects and adverse reactions of all patients will be observed and compared.

DETAILED DESCRIPTION:
According to strict inclusion and exclusion criteria, 99 newly diagnosed MM patients will be selected. They will be randomly assigned in a 2:1 ratio to the EAP group or the CG group. During the hematopoietic stem cell mobilization period, comparison study will be conducted regarding the proportion of patients who achieve the ideal collection value (CD34 cells >5×10^6/kg) after a single collection; the proportion of patients who cumulatively achieve the target collection value (CD34 cells >2×10^6/kg) and the ideal collection value; the cumulative collection of CD34 cells and the average number of collections; and the hematological and non-hematological adverse reactions of the EAP and CG regimens. Special attention will be given to the proportion of patients who add Plerixafor in both regimens.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients newly diagnosed as multiple myeloma.
* 2. Indication for ASCT.
* 3. Eastern Cooperative Oncology Group (ECOG) performance status of 0~1.
* 4. Life expectancy ≥ 3 months.
* 5. Subjects must be able to understand the protocol and sign the informed consent.

Exclusion Criteria:

* 1. Cardiac function class II or higher or cardiac ejection fraction <40%.
* 2. Serum direct bilirubin (DBIL)>2× upper limit of normal (ULN).
* 3. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3× ULN.
* 4. Serum creatinine clearance rate≤30%.
* 5. Patients with active infection.
* 6. Previously received hematopoietic stem cell mobilization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
% of patients achieving the collection of ≥5×10^6 CD34+ cells/kg | 1 month
  Proportion of patients who achieve the ideal collection value (CD34+ cells ≥5×10^6/kg) after a single collection

SECONDARY OUTCOMES:
% of patients achieving the collection of ≥2×10^6 CD34+ cells/kg | 1 month
  Comparison of the cumulative proportion of patients who achieve the target collection value (CD34+ cells ≥2×10^6/kg) between the EAP and CG regimens; the proportion of patients who achieve the ideal collection value.
CD34+ cells and the average number of collections | 1 month
  Comparison of the total amount of CD34+ cells collected and the average number of collections between the EAP and CG regimens.
Adverse Rvents (AEs) | 1 month
  Comparison of hematological and non-hematological adverse reactions between the EAP and CG regimens.
% of patients who use Plerixafor | 1 month
  Comparison of the proportion of patients who add Plerixafor between the EAP and CG regimens.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Lu, Principal Investigator — The Affiliated People's Hospital of Ningbo University
Locations (16):
- China (16):
  - Dongyang People's Hospital, Dongyang, Zhejiang
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Tongde Hospital of Zhejiang Province, Hangzhou, Zhejiang
  - Huzhou central hospital, Huzhou, Zhejiang
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang
  - Jinhua Municipal Central Hospital, Jinhua, Zhejiang
  - Jinhua People's Hospital, Jinhua, Zhejiang
  - Lishui Central Hospital, Lishui, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang
  - The Affiliated People's Hospital of Ningbo University, Ningbo, Zhejiang
  - Shaoxing People's Hospital, Shaoxing, Zhejiang
  - Shaoxing Second Hospital, Shaoxing, Zhejiang
  - Taizhou Central Hospital, Taizhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang